CLINICAL TRIAL: NCT01506986
Title: Helicobacter Eradication to Prevent Ulcer Bleeding in Aspirin Users: a Large Simple Randomised Controlled Trial
Brief Title: Helicobacter Eradication Aspirin Trial
Acronym: HEAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); University of Southampton (Other); University of Durham (Other); University of Birmingham (Other); University of Oxford (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11091; 09/55/52 (Other Grant/Funding Number: NIHR HTA); 2011-003425-96 (EudraCT Number); ISRCTN10134725 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Gastrointestinal Ulcer Haemorrhage; Bacterial Infection Due to Helicobacter Pylori (H. Pylori)
Keywords: Ulcer bleeding; Aspirin; Helicobacter pylori; H. pylori; Hospitalisation for ulcer bleeding
MeSH Terms: interventions — Lansoprazole; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H. pylori eradication treatment (Active Comparator): Active treatment will consist of seven days of lansoprazole 30mg twice daily, clarithromycin 500mg twice daily and metronidazole 400mg twice daily.
  Interventions: Drug: Lansoprazole 30mg, Clarithromycin 500mg, Metronidazole 400mg
- Placebo H. pylori eradication treatment (Placebo Comparator): Placebos to seven days of lansoprazole 30mg twice daily, clarithromycin 500mg twice daily and metronidazole 400mg twice daily.
  Interventions: Drug: Placebo lansoprazole 30mg, clarithromycin 500mg, metronidazole 400mg

INTERVENTIONS:
Drug: Lansoprazole 30mg, Clarithromycin 500mg, Metronidazole 400mg — All three medications will be taken orally, twice daily, for seven days.
  Other Names: Lansoprazole (CAS: 103577-45-3); 30mg capsules.; Clarithromycin (CAS: 81103-11-9); 500mg tablets.; Metronidazole (CAS: 99616-64-5) 400mg tablets.
  Arms: H. pylori eradication treatment
Drug: Placebo lansoprazole 30mg, clarithromycin 500mg, metronidazole 400mg — Medication to be taken orally, twice a day, for seven days.
  Arms: Placebo H. pylori eradication treatment

SUMMARY:
HEAT (Helicobacter Eradication Aspirin Trial) is a large simple double-blind placebo controlled outcomes study of Helicobacter pylori (H. pylori) eradication to prevent ulcer bleeding in aspirin users. It will be run by the University of Nottingham, with recruiting centres across the UK. This trial is funded by the National Institute of Health Research Health Technology Assessment (NIHR HTA) Programme.

Aspirin use is widespread and increasing in elderly patients. The main hazard is gastrointestinal bleeding, which may be increasing because of increasing aspirin use. This trial is based on evidence that peptic ulcer bleeding in aspirin users occurs predominantly in H. pylori positive people.

Patients will be identified by their GPs, then asked to attend an appointment with a Research Nurse to consent to the trial and take a H. pylori breath test. Those with a positive result will be randomised to receive a one week course of either eradication treatment or placebo. No follow-up visits are required, but instead information will be extracted from the patients' electronic medical record using the MiQuest search tool.

The trial will continue until 87 adjudicated events (hospitalisation because of definite or probable peptic ulcer bleeding) have occurred, which would occur after a mean 2.5 patient years of follow-up, if trial assumptions are correct.

DETAILED DESCRIPTION:
BACKGROUND: Aspirin use is widespread and increasing in elderly patients. The main hazard is gastrointestinal bleeding, the incidence of which is rising, probably because of increased aspirin use. The proposed trial is based on evidence that peptic ulcer bleeding in aspirin users occurs predominantly in people infected with the ulcerogenic bacterium, Helicobacter pylori. Our hypothesis is that low doses of aspirin do not cause ulcers in the way that high doses do. Instead we think that H. pylori causes the ulcer and aspirin, by thinning the blood, makes it bleed. If the bacterium is eradicated the patient will not get an ulcer and therefore there is no increased bleeding risk with aspirin. Development of the trial protocol has been based on results of a preparatory Medical Research Council-funded 2525 patient pilot study which had a 47% patient response rate. This enabled us to design the currently proposed large simple outcomes study to investigate directly the hypothesis that a one week course of H. pylori eradication will halve the rate of hospitalisation due to ulcer bleeding over ~2.5 years in aspirin users.

TRIAL CONDUCT: A large number of patients (~170,000), using aspirin <326 mg daily will be invited to participate. Suitable respondents (~33,000) who are H. pylori positive (~6,600) will give consent (including access to Hospital Episode Statistics and Office of National Statistics mortality data) and be randomised to eradication treatment or placebo. There will be no follow-up trial visits for 90% of patients. Instead the MiQuest tool, developed to interrogate different GP electronic databases, will be used together with direct patient notification to identify all possible ulcer bleeding admissions. An expert panel will use validated methodology to adjudicate whether patients have suffered ulcer bleeding (primary endpoint). The trial will continue until 87 positively adjudicated events have occurred, to ensure it has the power to answer the question of whether H. pylori eradication reduces the risk of ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 60 years of age at the date of screening.
* Subjects who are taking aspirin ≤325mg daily and who have had 4 or more 28-day prescriptions in the last year.
* Subjects who are concurrently using other anti-platelet agents are allowed to enter the study.
* Subjects who are willing and able to undergo a breath test for H. pylori, including fasting for 6 hours, and whose result is unequivocally positive (results of breath test will be determined post-screening).
* Subjects who are willing to give permission for their paper and electronic medical records to be accessed and abstracted by trial investigators.
* Subjects who are willing to be contacted and interviewed by trial investigators, should the need arise for adverse event assessment, etc.
* Subjects must be able to communicate well with the investigator or designee, to understand and comply with the requirements of the study and to understand and sign the written informed consent.

Exclusion Criteria:

* Subjects who are currently prescribed anti-ulcer therapy such as H2-receptor antagonists and proton-pump inhibitors.
* Subjects who are currently prescribed oral non-steroidal anti-inflammatory drugs (NSAIDs).
* Subjects who have a known intolerance or allergy to H. pylori eradication treatment.
* Subjects who are taking drugs with a clinically significant interaction with H. pylori eradication treatment.
* Subjects who are terminally ill or suffer from a life-threatening co-morbidity.
* Subjects whose behaviour or lifestyle would render them less likely to comply with study medication (eg. alcoholism, substance abuse, debilitating psychiatric conditions or inability to provide informed consent).
* Subjects currently participating in another interventional clinical trial or who have taken part in a trial in the previous three months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30024 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
The rate of hospitalisation due to peptic ulcer bleeding in patients who enter the randomised study (only the first event per patient will be analysed), adjudicated by a blinded Committee as definite or probable. | 4 years

SECONDARY OUTCOMES:
Other causes of gastrointestinal bleeding (adjudicated); these are predicted not to be affected by H. pylori eradication and will act as a specificity control. | 4 years
Cardiovascular outcomes (APTC (Anti Platelet Trialists Collaboration) endpoint, myocardial infarction and stroke, unadjudicated); these are predicted not to be affected. | 4 years
The incidence of detected uncomplicated ulcers. | 4 years
Ulcer site (Duodenal Ulcer vs. Gastric Ulcer). | 4 years
GP-recorded and patient-reported dyspepsia. | 4 years
Need for proton pump inhibitor prescription or other antiulcer/dyspepsia medication. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Chris J Hawkey, Principal Investigator — University of Nottingham
Locations (6):
- United Kingdom (6):
  - Queen's University, Belfast
  - University of Birmingham, Birmingham
  - Durham University, Durham
  - University of Nottingham, Nottingham
  - University of Oxford, Oxford
  - University of Southampton, Southampton

REFERENCES:
- [Background] Dumbleton JS, Avery AJ, Coupland C, Hobbs FD, Kendrick D, Moore MV, Morris C, Rubin GP, Smith MD, Stevenson DJ, Hawkey CJ. The Helicobacter Eradication Aspirin Trial (HEAT): A Large Simple Randomised Controlled Trial Using Novel Methodology in Primary Care. EBioMedicine. 2015 Jul 10;2(9):1200-4. doi: 10.1016/j.ebiom.2015.07.012. eCollection 2015 Sep. PMID 26501118
- [Derived] Hawkey CJ, Avery AJ, Coupland CA, Crooks CJ, Dumbleton JS, Hobbs FR, Kendrick D, Moore M, Morris C, Rubin G, Smith M, Stevenson D; HEAT trialists. Eradication of Helicobacter pylori for prevention of aspirin-associated peptic ulcer bleeding in adults over 65 years: the HEAT RCT. Health Technol Assess. 2025 Aug;29(42):1-62. doi: 10.3310/LLKF7871. PMID 40844182
- [Derived] Stevenson DJ, Avery AJ, Coupland C, Hobbs FDR, Kendrick D, Moore MV, Morris C, Rubin GP, Smith MD, Hawkey CJ, Dumbleton JS. Recruitment to a large scale randomised controlled clinical trial in primary care: the Helicobacter Eradication Aspirin Trial (HEAT). Trials. 2022 Feb 14;23(1):140. doi: 10.1186/s13063-022-06054-w. PMID 35164864